CLINICAL TRIAL: NCT00603187
Title: Oral Administration of the GnRH Antagonist Acyline in Normal Men Part II: Multiple-dose Pharmacokinetics (Acyline-7/MER 104-02)
Brief Title: ACY-7 Oral Administration of Acyline
Acronym: ACY-7
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Merrion Pharmaceuticals, LLC (Industry)
Responsible Party: John K Amory, MD, MPH, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 32716-W; 07-7973-W (Other: UW Human Subjects Division)
Record Dates: First submitted 2008-01-15; First posted 2008-01-28 (Estimated); Results first posted 2011-06-09 (Estimated); Last update posted 2011-06-09 (Estimated); Status verified 2011-05

CONDITIONS: Healthy
Keywords: Male Contraception; Acyline
MeSH Terms: interventions — acyline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Acyline — 20 mg GIPET enhanced oral dose, daily for 7-days

SUMMARY:
We propose oral dosing of gastrointestinal permeation enhancement technology [GIPET] enhanced oral acyline at 20 mg everyday for one week to determine the steady-state (multiple-dose) pharmacokinetics of oral acyline in four normal, healthy young men.

DETAILED DESCRIPTION:
The purpose of this study is to test how the body responds to a new oral form of acyline given for seven days and to also look at the safety of oral acyline.

Acyline temporarily blocks the production of the hormone testosterone in healthy men. It has been tested in over 100 men in an injection form. This study will be testing acyline in a pill form for seven days.

This study may help develop an oral form of testosterone-blocker which may be useful in the treatment of diseases such as prostate cancer, premature puberty and possibly in a male contraceptive.

This study will evaluate a single dose of oral acyline given once a day for seven days and subsequent effects on Testosterone, FSH and LH blood serum concentrations.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male
* 18-50 years of age
* Non-smoker
* Not taking any medications other than the study drug for the duration of the study.
* Must be willing to use an accepted method of contraception during the study.

Exclusion Criteria:

* BMI > 35
* Abnormal evaluation on screening exam and labs
* Known history of alcohol abuse, illicit drugs or steroids and/or use of more that 3 alcoholic beverages/day
* History of current testosterone use or infertility
* History of testicular disease or severe testicular trauma
* History of major psychiatric disorder or sleep apnea
* History of bleeding disorder or need for anticoagulation
* Current smoker or utilizing nicotine patches or gum
* Participation in a hormonal drug study within past month.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2008-01; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John K Amory, MD, MPH, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

REFERENCES:
- [Background] Herbst KL, Anawalt BD, Amory JK, Bremner WJ. Acyline: the first study in humans of a potent, new gonadotropin-releasing hormone antagonist. J Clin Endocrinol Metab. 2002 Jul;87(7):3215-20. doi: 10.1210/jcem.87.7.8675. PMID 12107227
- [Background] Herbst KL, Coviello AD, Page S, Amory JK, Anawalt BD, Bremner WJ. A single dose of the potent gonadotropin-releasing hormone antagonist acyline suppresses gonadotropins and testosterone for 2 weeks in healthy young men. J Clin Endocrinol Metab. 2004 Dec;89(12):5959-65. doi: 10.1210/jc.2003-032123. PMID 15579744
- [Background] Matthiesson KL, Amory JK, Berger R, Ugoni A, McLachlan RI, Bremner WJ. Novel male hormonal contraceptive combinations: the hormonal and spermatogenic effects of testosterone and levonorgestrel combined with a 5alpha-reductase inhibitor or gonadotropin-releasing hormone antagonist. J Clin Endocrinol Metab. 2005 Jan;90(1):91-7. doi: 10.1210/jc.2004-1228. Epub 2004 Oct 27. PMID 15509637
- [Background] Amory JK, Bremner WJ. Oral testosterone in oil plus dutasteride in men: a pharmacokinetic study. J Clin Endocrinol Metab. 2005 May;90(5):2610-7. doi: 10.1210/jc.2004-1221. Epub 2005 Feb 15. PMID 15713724
- [Background] Amory JK, Page ST, Bremner WJ. Oral testosterone in oil: pharmacokinetic effects of 5alpha reduction by finasteride or dutasteride and food intake in men. J Androl. 2006 Jan-Feb;27(1):72-8. doi: 10.2164/jandrol.05058. PMID 16400081
- [Background] Page ST, Lin DW, Mostaghel EA, Hess DL, True LD, Amory JK, Nelson PS, Matsumoto AM, Bremner WJ. Persistent intraprostatic androgen concentrations after medical castration in healthy men. J Clin Endocrinol Metab. 2006 Oct;91(10):3850-6. doi: 10.1210/jc.2006-0968. Epub 2006 Aug 1. PMID 16882745
- [Background] Page ST, Amory JK, Anawalt BD, Irwig MS, Brockenbrough AT, Matsumoto AM, Bremner WJ. Testosterone gel combined with depomedroxyprogesterone acetate is an effective male hormonal contraceptive regimen and is not enhanced by the addition of a GnRH antagonist. J Clin Endocrinol Metab. 2006 Nov;91(11):4374-80. doi: 10.1210/jc.2006-1411. Epub 2006 Aug 29. PMID 16940442

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited via fliers on the University of Washington campus.
Pre-assignment Details: Healthy, non-smoking male subjects between 18-50 years of age were recruited. Health was determined by physical exam, medical history intake and laboratory blood tests.
Groups:
- Oral Acyline: 20 mg dose of GIPET enhanced oral acyline for 7 days
Period: Overall Study
Arm/Group | Oral Acyline
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Oral Acyline
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 40 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Testosterone Blood Serum Concentration
Description: Blood for measurement of serum testosterone was obtained prior to the 1st, 5th and 6th dose of GIPET™-enhanced oral acyline and 0.5,1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48 and 60 hours after the 7th dose.
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: ng/dl
Arm/Group | Oral Acyline
Number analyzed (Participants) | 4
ng/dl
  pre-dose 1 | 14.25 (4.72)
  pre-dose 5 | 8.53 (2.06)
  pre-dose 6 | 9.83 (1.93)
  pre-dose 7 | 9.83 (3.39)
  dose 7, 0.5 hours | 10.10 (3.73)
  dose 7, 1 hour | 9.50 (3.67)
  dose 7, 1.5 hours | 10.33 (4.35)
  dose 7, 2 hours | 10.65 (3.38)
  dose 7, 3 hours | 9.80 (4.05)
  dose 7, 4 hours | 8.78 (3.18)
  dose 7, 6 hours | 7.08 (2.84)
  dose 7, 8 hours | 6.80 (3.70)
  dose 7, 12 hours | 6.88 (3.81)
  dose 7, 24 hours | 9.30 (4.58)
  dose 7, 36 hours | 8.20 (2.71)
  dose 7, 48 hours | 10.83 (4.29)
  dose 7, 60 hours | 10.10 (4.61)
  Recovery/day 14 | 16.5 (2.12)

2. Secondary Outcome: FSH Blood Serum Concentration
Description: Blood for measurement of serum follicle stimulating hormone concentrations was obtained prior to the 1st, 5th and 6th dose of GIPET™-enhanced oral acyline and 0.5,1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48 and 60 hours after the 7th dose.
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: iu/L
Arm/Group | Oral Acyline
Number analyzed (Participants) | 4
iu/L
  pre-dose 1 | 2.80 (1.55)
  pre-dose 5 | 2.05 (0.60)
  pre-dose 6 | 2.33 (0.69)
  pre-dose 7 | 2.23 (0.72)
  dose 7, 0.5 hours | 2.48 (0.67)
  dose 7, 1 hour | 2.38 (0.69)
  dose 7, 1.5 hours | 2.45 (0.83)
  dose 7, 2 hours | 2.45 (0.77)
  dose 7, 3 hours | 2.33 (0.78)
  dose 7, 4 hours | 2.20 (0.92)
  dose 7, 6 hours | 2.05 (0.61)
  dose 7, 8 hours | 1.93 (0.62)
  dose 7, 12 hours | 2.03 (0.59)
  dose 7, 24 hours | 2.28 (0.62)
  dose 7, 36 hours | 2.48 (0.85)
  dose 7, 48 hours | 3.00 (1.11)
  dose 7, 60 hours | 2.93 (1.21)
  Recovery/day 14 | 3.20 (2.83)

3. Secondary Outcome: LH Blood Serum Concentration
Description: Blood for measurement of serum leutenizing hormone concentrations was obtained prior to the 1st, 5th and 6th dose of GIPET™-enhanced oral acyline and 0.5,1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48 and 60 hours after the 7th dose.
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: iu/L
Arm/Group | Oral Acyline
Number analyzed (Participants) | 4
iu/L
  pre-dose 1 | 4.87 (5.53)
  pre-dose 5 | 2.73 (1.53)
  pre-dose 6 | 4.78 (4.43)
  pre-dose 7 | 4.15 (4.60)
  dose 7, 0.5 hours | 5.80 (2.82)
  dose 7, 1 hour | 5.18 (3.90)
  dose 7, 1.5 hours | 5.30 (5.15)
  dose 7, 2 hours | 5.40 (4.56)
  dose 7, 3 hours | 3.83 (3.35)
  dose 7, 4 hours | 2.98 (2.67)
  dose 7, 6 hours | 2.35 (1.66)
  dose 7, 8 hours | 1.94 (1.46)
  dose 7, 12 hours | 2.40 (1.25)
  dose 7, 24 hours | 4.10 (2.68)
  dose 7, 36 hours | 6.70 (6.21)
  dose 7, 48 hours | 7.20 (7.88)
  dose 7, 60 hours | 5.80 (6.25)
  Recovery/day 14 | 8.10 (9.76)

ADVERSE EVENTS:
Arm/Group | Oral Acyline
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No